CLINICAL TRIAL: NCT05847010
Title: Accompanying Scientific Program for the Quality Contract Prevention of Postoperative Delirium in the Care of Older Patients (WB-QC-POD)
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiolgy and Intensive Care Medicine CC07, Charite University, Berlin, Germany
Other Study IDs: WB-QC-POD
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (monocytes and Cholinesterase activity)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the course of a scientific accompanying program, the project pursues the goal of gaining further insight into a possible connection between various influencing factors and the development of postoperative delirium. Against this background, in addition to the primary goal of exploring delirium rates, we aim to identify associations between other secondary end goals like the internal circadian time or the heart rate variability and the occurrence of postoperative delirium. For this purpose, patients of the QC-POD (NCT04355195) sample will be studied.

DETAILED DESCRIPTION:
The project aims to improve the understanding of the internal circadian time (chronotype) and other sleep parameters, as well as further secondary end goals, in relation to the development of postoperative delirium. In the course of this the project would like to investigate the perioperative heart rate variability. Also, the association of perioperative peripheral cholinesterase activity with perioperative heart rate variability and the development of POD will be explored. Additionally, the investigator will analyze the correlation of intraoperative EEG signatures with perioperative heart rate variability, and explore any association of core body temperature and the development of postoperative Delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Male and female patients
* Patients who have been included in QC-POD
* Eligible patients* for inclusion: informed consent by the patient, preoperatively with verbal and written informed consent before the start of data collection
* Incapacitated patients for inclusion: Written informed consent by a legal representative
* surgery (elective and not elective)

Exclusion Criteria:

* Moribund patients (palliative situation)
* Insufficient knowledge of the German language
* Cardiac arrhythmia (e.g. atrial fibrillation)
* Presence of a pacemaker
* Condition after heart transplantation
* Inflammation in the area of the frontal sinus

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥70 years, male and female, who are receiving surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative Delirium | Up to the fifth postoperative day
  Incidence of postoperative delirium in all postoperative patients in normal ward, intensive care unit and recovery room with a validated delirium screening tool at two points in time.

SECONDARY OUTCOMES:
Duration of Delirium | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Duration (in days) of postoperative delirium in all postoperative patients in normal ward, intensive care unit and recovery room with a validated delirium screening tool at two points in time.
Bodytime | Before surgery
  Bodytime is determined from monocytes on the morning of surgery.
Chronotype 1 | Up to three months
  "Munich ChronoType Questionnaire" (MCTQ), modified for seniors is measured preoperatively and 3 months postoperatively
Chronotype 2 | Up to three months
  "Morningness-Eveningness-Questionnaire" (D-MEQ) is measured preoperatively and 3 months postoperatively
Heart rate variability 1 | The participants are followed up until the end of hospital stay, an expected average of 7 days.
  Heartrate variability 1 is measured by "ANI Monitor V2" until discharge. With the "Ani Monitor V2", heart rate variability is recorded twice a day and intraoperatively.
Heart rate variability 2 | The participants are followed up until the end of hospital stay, an expected average of 7 days.
  Heartrate variability 2 is measured by "Bittium Faros 180" until discharge, except during surgery.
Body core temperature | Up to the third postoperative day
  Body core temperature is measured with "Tcore™", a new non-invasive technology, which employs a unique dual-sensor heat flux technology.
Electroencephalography signatures | During surgery, an expected time of two hours.
  Electroencephalography signatures are measured during surgery.
Sleep monitoring 1 | Up to the third postoperative day
  Sleep should be measured with a "Sleep Profiler" that generates electrooculography data.
Sleep monitoring 2 | Up to the third postoperative day
  Sleep should be measured with a "Sleep Profiler" that generates electroencephalography data.
Sleep monitoring 3 | Up to the third postoperative day
  Sleep should be measured with a "Sleep Profiler" that generates electromyogram data.
Insomnia Severity Index | Up to three months
  Patients will assess their sleep quality by Insomnia Severity Index questionnaire.

OTHER OUTCOMES:
Proteomics | At the morning of surgery
  Biomarkers of delirium based on proteomics, measured by analysis of a plasma sample.
Metabolomics | At the morning of surgery
  Biomarkers of delirium based on metabolomics, measured by analysis of a plasma sample.
Bodytime | At the morning of surgery
  Biomarkers of chrono type based on body time, measured by analysis of monocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum (CVK) and Campus Charite Mitte (CCM), Charite - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No